CLINICAL TRIAL: NCT05175638
Title: Macrophage Migration Inhibiting Factor, Enolase and Caspase-3 as Indicators of Neuronal Insult in Newborns of COVID-19 Positive Mothers.
Brief Title: Indicators of Neuronal Insult in Newborns of COVID-19 Positive Mothers.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Mohammed Ali, Principal investigator, Assiut University
Other Study IDs: NER
Record Dates: First submitted 2022-01-01; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — Gene Expression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: A total of 20 term newborn infants with a median gestational age of 40 weeks (range: 37-42 weeks) will be selected from the Gynecology and Obstetrics Hospital (Assiut University). All control infants should have an Apgar score of > 9 at 1, 5, and 10 minutes.
  Interventions: Genetic: Gene Expression
- Study group: Thirty newborn infants born for Covid-19 positive mothers will be prospectively included in this study. The diagnosis of hypoxia will made based on Apgar score, clinical signs present during the first hours of life and acid-base status.
  The following inclusion criteria will be used (all necessary): Covid-19 positive mothers, term newborn (>37 completed gestational weeks), free from severe malformations. All infants will be examined generally, systemically and neurologically at birth for clinical assessment of HIE if present and for detection of outcome of these neonates.
  Interventions: Genetic: Gene Expression

INTERVENTIONS:
Genetic: Gene Expression — the expression of specific CNS enzyme (enolase), proinflammatory cytokines MIF and apoptotic marker caspase-3 in the umbilical blood of infants delivered for Covid positive mothers.

SUMMARY:
The coronavirus disease (COVID- 19) is now a global pandemic that was first reported in China (Wuhan) in December of 2019. Multiple placental abnormalities including fetal and maternal vascular malperfusion have been described in pregnant women infected with (COVID- 19). To date, there are far fewer reports about the specific effects of (COVID- 19) in the newborns delivered for (COVID- 19) positive mothers.

DETAILED DESCRIPTION:
COVID-19 in pregnant women has important impacts on perinatal and neonatal outcomes. Authors reported positive COVID infection in neonates born to COVID-19 positive mother.

The finding of a recent study suggested that intrauterine or intrapartum transmission is possible and recommended for further investigation. Furthermore, reports showed newborns of COVID-19 positive mother that suffered from catastrophic sequelae of hypoxic ischemic encephalopathy (HIE). These events could be attributed to COVID-19 positive status of the mother.

Neuron specific enolase is a biomarker for neuronal injury and synaptic dysfunction and have been correlated with tissue damage in different experimental models. The increased serum levels of neuron specific enolase are associated with the clinical outcome in patients with anoxic encephalopathy. Neuron specific enolase can be a candidate for a diagnostic/prognostic biomarker for neuroinflammation in COVID-19.

Additionally, the cytokines are candidate biomarkers after hypoxic-ischemic injury. Macrophage migration inhibitory factor (MIF) is a multifunctional protein that has been identified as proinflammatory cytokine and activates the production of inflammatory cytokines such as tumor necrosis factor-α, interleukin-1β, interleukin-6, and interferon.

Macrophage migration inhibitory factor plays a central role in controlling the inflammatory and immune response, which may be of particular importance during the development of organ dysfunction in COVID-19 patients. Furthermore, it carries out the apoptosis of the cells. Significant increase of neuronal apoptosis and caspase-3 expression was demonstrated in the brain of neonatal mice exposed to hypoxic injury.

There are a limited number of studies investigating the effect of the pandemic period on the brain of the newborns. With this study, we aim to determine the impact of the COVID-19 outbreak on the neuronal functions in the neonates. The current study searches for a diagnostic/prognostic biomarker for neuroinflammation in neonate born to COVID-19 positive mothers.

ELIGIBILITY:
Inclusion Criteria:

* The following inclusion criteria will be used (all necessary): Covid-19 positive mothers, term newborn (>37 completed gestational weeks), free from severe malformations. All infants will be examined generally, systemically and neurologically at birth for clinical assessment of HIE if present and for detection of outcome of these neonates.

Exclusion Criteria:

* free from severe malformations

Ages: 1 Day to 2 Days | Sex: All
Age Groups: Child
Study Population: Fifty newborn babies will be recruited from Assiut university hospital and included in this study. Thirty newborn babies delivered for COVID 19 positive mothers, and 20 newborns delivered for normal mothers will be used as control group. Informed consent will be obtained from mothers.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
the expression of specific CNS enzyme (enolase), proinflammatory cytokines MIF and apoptotic marker caspase-3 in the umbilical blood of infants delivered for Covid positive mothers. | one month
  RNA extraction Reverse Transcription polymerase chain reaction (RT-PCR) analysis:

REFERENCES:
- [Background] Aksakal A, Kerget B, Kerget F, Askin S. Evaluation of the relationship between macrophage migration inhibitory factor level and clinical course in patients with COVID-19 pneumonia. J Med Virol. 2021 Dec;93(12):6519-6524. doi: 10.1002/jmv.27189. Epub 2021 Jul 22. PMID 34241898
- [Background] Bleilevens C, Soppert J, Hoffmann A, Breuer T, Bernhagen J, Martin L, Stiehler L, Marx G, Dreher M, Stoppe C, Simon TP. Macrophage Migration Inhibitory Factor (MIF) Plasma Concentration in Critically Ill COVID-19 Patients: A Prospective Observational Study. Diagnostics (Basel). 2021 Feb 17;11(2):332. doi: 10.3390/diagnostics11020332. PMID 33671433
- [Background] Chaparro-Huerta V, Flores-Soto ME, Merin Sigala ME, Barrera de Leon JC, Lemus-Varela ML, Torres-Mendoza BM, Beas-Zarate C. Proinflammatory Cytokines, Enolase and S-100 as Early Biochemical Indicators of Hypoxic-Ischemic Encephalopathy Following Perinatal Asphyxia in Newborns. Pediatr Neonatol. 2017 Feb;58(1):70-76. doi: 10.1016/j.pedneo.2016.05.001. Epub 2016 May 31. PMID 27522459
- [Background] Deng C, Li J, Li L, Sun F, Xie J. Effects of hypoxia ischemia on caspase-3 expression and neuronal apoptosis in the brain of neonatal mice. Exp Ther Med. 2019 Jun;17(6):4517-4521. doi: 10.3892/etm.2019.7487. Epub 2019 Apr 15. PMID 31086583
- [Background] Florez-Sampedro L, Brandsma CA, de Vries M, Timens W, Bults R, Vermeulen CJ, van den Berge M, Obeidat M, Joubert P, Nickle DC, Poelarends GJ, Faiz A, Melgert BN. Genetic regulation of gene expression of MIF family members in lung tissue. Sci Rep. 2020 Oct 12;10(1):16980. doi: 10.1038/s41598-020-74121-w. PMID 33046825
- [Background] Ganti L, Serrano E, Toklu HZ. Can Neuron Specific Enolase Be a Diagnostic Biomarker for Neuronal Injury in COVID-19? Cureus. 2020 Oct 19;12(10):e11033. doi: 10.7759/cureus.11033. PMID 33214960
- [Background] Gladkevich A, Kauffman HF, Korf J. Lymphocytes as a neural probe: potential for studying psychiatric disorders. Prog Neuropsychopharmacol Biol Psychiatry. 2004 May;28(3):559-76. doi: 10.1016/j.pnpbp.2004.01.009. PMID 15093964
- [Background] Golden TN, Simmons RA. Maternal and neonatal response to COVID-19. Am J Physiol Endocrinol Metab. 2020 Aug 1;319(2):E315-E319. doi: 10.1152/ajpendo.00287.2020. Epub 2020 Jun 23. PMID 32574110
- [Background] Haque A, Polcyn R, Matzelle D, Banik NL. New Insights into the Role of Neuron-Specific Enolase in Neuro-Inflammation, Neurodegeneration, and Neuroprotection. Brain Sci. 2018 Feb 18;8(2):33. doi: 10.3390/brainsci8020033. PMID 29463007
- [Background] Hekimoglu B, Akturk Acar F. Effects of COVID-19 pandemic period on neonatal mortality and morbidity. Pediatr Neonatol. 2022 Jan;63(1):78-83. doi: 10.1016/j.pedneo.2021.08.019. Epub 2021 Oct 27. PMID 34776364
- [Background] Isgro MA, Bottoni P, Scatena R. Neuron-Specific Enolase as a Biomarker: Biochemical and Clinical Aspects. Adv Exp Med Biol. 2015;867:125-43. doi: 10.1007/978-94-017-7215-0_9. PMID 26530364
- [Background] Jain P, Thakur A, Kler N, Garg P. Manifestations in Neonates Born to COVID-19 Positive Mothers. Indian J Pediatr. 2020 Aug;87(8):644. doi: 10.1007/s12098-020-03369-x. Epub 2020 Jun 5. No abstract available. PMID 32504454
- [Background] Wang S, Guo L, Chen L, Liu W, Cao Y, Zhang J, Feng L. A Case Report of Neonatal 2019 Coronavirus Disease in China. Clin Infect Dis. 2020 Jul 28;71(15):853-857. doi: 10.1093/cid/ciaa225. PMID 32161941
- [Background] Wu YT, Liu J, Xu JJ, Chen YF, Yang W, Chen Y, Li C, Wang Y, Liu H, Zhang C, Jiang L, Qian ZX, Kawai A, Mol BW, Dennis CL, Xiong GP, Cheng BH, Yang J, Huang HF. Neonatal outcome in 29 pregnant women with COVID-19: A retrospective study in Wuhan, China. PLoS Med. 2020 Jul 28;17(7):e1003195. doi: 10.1371/journal.pmed.1003195. eCollection 2020 Jul. PMID 32722722
- [Background] Zeng L, Xia S, Yuan W, Yan K, Xiao F, Shao J, Zhou W. Neonatal Early-Onset Infection With SARS-CoV-2 in 33 Neonates Born to Mothers With COVID-19 in Wuhan, China. JAMA Pediatr. 2020 Jul 1;174(7):722-725. doi: 10.1001/jamapediatrics.2020.0878. PMID 32215598